CLINICAL TRIAL: NCT04342091
Title: Follicular Revival in Fibrosing Alopecia: Evaluating Use of Micro-needling
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2000027405
Record Dates: First submitted 2020-04-06; First posted 2020-04-10 (Actual); Results first posted 2023-04-13 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-03

CONDITIONS: Fibrosing Alopecia; Frontal Fibrosing Alopecia; Central Centrifugal Cicatricial Alopecia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Microneedling (Experimental): Participants with fibrosing alopecia will receive microneedling with a tattoo machine.
  Interventions: Device: SOL Nova Device

INTERVENTIONS:
Device: SOL Nova Device — A SOL Nova Device (brand) is tattoo machine will be used to stimulate hair regrowth.

SUMMARY:
To evaluate the efficacy microneedling via a professional tattoo machine in revitalizing hair follicles in patients with fibrosing alopecia.

DETAILED DESCRIPTION:
The investigators propose an open label trial of tattoo machine microneedling in ten patients with fibrosing alopecia (five patients with CCCA and five with FFA). Ten healthy female patients older than 18 years will undergo 6 microneedling sessions. Over the course of six months, subjects will undergo up to six treatment sessions (one session every 30 day). Photographs will be taken at each session. Patients will be evaluated at 8 visits over 8 months with the first visit for screening purposes. Each visit will last about an hour. Approximately 30 minutes will be spent on consenting and time for patient to ask questions during the first visit. The remaining 30 minutes will be allotted for the investigator to determine if the patient meets criteria for trial enrollment. During the remaining visits, 20 minutes will be allotted for photography, 15-20 minutes for the procedure and 10-15 minutes for post-procedure patient assessment. Remaining 10 minutes on visits 2 and 8 will be used for biopsy.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Female
* Diagnosing Fibrosing alopecia

Exclusion Criteria:

* Any female with hair loss for other reasons
* Males
* Patients with cardiac conditions or renal insufficiency
* Pregnant patients
* Patients containing the following who would make poor candidates for microneedling, such as skin conditions, diabetes, history of keloid formation
* Anything additional existing comorbidities that in the opinion of the investigator may cause unnecessary risk for the patient to participate

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2021-04-09 (Actual); Primary Completion 2022-04-08 (Actual); Study Completion 2022-04-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brett King, MD, PhD, Principal Investigator — Associate Professor of Dermatology, Yale University
Locations (1):
- Yale University, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Microneedling
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Microneedling
Number analyzed (Participants) | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.8 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Total area hair count (frontal) [Mean (Standard Deviation); unit: Count per cm^2] — Population: 4 participants with frontal area analyzed (area of involvement)
  Count per cm^2
    number analyzed (Participants) | 4
    (all) | 50.0 (66.3)
Total hair count (vertex) [Mean (Standard Deviation); unit: Count per cm^2] — Population: 2 participants with vertex area analyzed (area of involvement)
  Count per cm^2
    number analyzed (Participants) | 2
    (all) | 32.5 (6.4)
Hair shaft diameter (frontal) [Mean (Standard Deviation); unit: micrometer] — Population: 4 participants with frontal area analyzed (area of involvement)
  micrometer
    number analyzed (Participants) | 4
    (all) | 62.3 (16.5)
Hair shaft diameter (vertex) [Mean (Standard Deviation); unit: micrometer] — Population: 2 participants with vertex area analyzed (area of involvement)
  micrometer
    number analyzed (Participants) | 2
    (all) | 72.2 (7.1)
Number of hair follicles (frontal) [Mean (Standard Deviation); unit: follicle count per cm^2] — Population: 4 participants with frontal area analyzed (area of involvement)
  follicle count per cm^2
    number analyzed (Participants) | 4
    (all) | 46.0 (55.8)
Number of hair follicles (vertex) [Mean (Standard Deviation); unit: follicle count per cm^2] — Population: 2 participants with vertex area analyzed (area of involvement)
  follicle count per cm^2
    number analyzed (Participants) | 2
    (all) | 31.5 (2.1)
Vellus hairs (frontal) [Mean (Standard Deviation); unit: Count per cm^2] — Population: 4 participants with frontal area analyzed (area of involvement)
  Count per cm^2
    number analyzed (Participants) | 4
    (all) | 0.8 (1.5)
Vellus hairs (vertex) [Mean (Standard Deviation); unit: Count per cm^2] — Population: 2 participants with vertex area analyzed (area of involvement)
  Count per cm^2
    number analyzed (Participants) | 2
    (all) | 0 (0)
Terminal hairs (frontal) [Mean (Standard Deviation); unit: Count per cm^2] — Population: 4 participants with frontal area analyzed (area of involvement)
  Count per cm^2
    number analyzed (Participants) | 4
    (all) | 49.3 (66.8)
Terminal hairs (vertex) [Mean (Standard Deviation); unit: Count per cm^2] — Population: 2 participants with vertex area analyzed (area of involvement)
  Count per cm^2
    number analyzed (Participants) | 2
    (all) | 32.5 (6.4)

OUTCOME MEASURES:

1. Primary Outcome: Total Area Hair Count (Frontal)
Description: Total number of hairs over an area of 1cm^2
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: Count per cm^2
Arm/Group | Microneedling
Number analyzed (Participants) | 4
Count per cm^2 | 86.8 (73.0)

2. Primary Outcome: Total Area Hair Count (Vertex)
Description: Total number of hairs over an area of 1 cm^2
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: Count per cm^2
Arm/Group | Microneedling
Number analyzed (Participants) | 2
Count per cm^2 | 117.5 (115.3)

3. Secondary Outcome: Hair Shaft Diameters (Frontal)
Description: Hair shaft diameter measured per trichoscopy
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: micrometer
Arm/Group | Microneedling
Number analyzed (Participants) | 4
micrometer | 61.1 (19.6)

4. Secondary Outcome: Hair Shaft Diameters (Vertex)
Description: Hair shaft diameter measured per trichoscopy
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: micrometer
Arm/Group | Microneedling
Number analyzed (Participants) | 2
micrometer | 63.5 (5.2)

5. Secondary Outcome: Number of Hair Follicles (Frontal)
Description: Number of hair follicles counted per 1cm^2
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: Count per cm^2
Arm/Group | Microneedling
Number analyzed (Participants) | 4
Count per cm^2 | 70.3 (59.6)

6. Secondary Outcome: Number of Hair Follicles (Vertex)
Description: Number of hair follicles per 1 cm^2
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: Count per cm^2
Arm/Group | Microneedling
Number analyzed (Participants) | 2
Count per cm^2 | 74.0 (53.7)

7. Secondary Outcome: Vellus Hairs (Frontal)
Description: Number of vellus hairs per cm^2
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: Count per cm^2
Arm/Group | Microneedling
Number analyzed (Participants) | 4
Count per cm^2 | 1.5 (3.0)

8. Secondary Outcome: Vellus Hairs (Vertex)
Description: Number of vellus hairs per cm^2
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: Count per cm^2
Arm/Group | Microneedling
Number analyzed (Participants) | 2
Count per cm^2 | 0 (0)

9. Secondary Outcome: Terminal Hairs (Frontal)
Description: Number of terminal hairs over an area of 1 cm^2
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: Count per cm^2
Arm/Group | Microneedling
Number analyzed (Participants) | 4
Count per cm^2 | 85.3 (74.6)

10. Secondary Outcome: Terminal Hairs (Vertex)
Description: Number of terminal hairs per area of 1 cm^2
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: Count per cm^2
Arm/Group | Microneedling
Number analyzed (Participants) | 2
Count per cm^2 | 117.5 (115.3)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Microneedling
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 2/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Microneedling (N=6)
Tongue Lesion (R Lateral Tongue) (Gastrointestinal disorders) | 1 (1)
Hair shedding (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-02): https://cdn.clinicaltrials.gov/large-docs/91/NCT04342091/Prot_SAP_000.pdf